CLINICAL TRIAL: NCT00908856
Title: Safety of IV Autologous Mononuclear Cells and Marrow Stromal Cells After Stroke
Brief Title: Autologous Cell Therapy After Stroke
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Not funded
Sponsor: University of California, Irvine (Other)
Collaborators: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Steven C. Cramer, MD, Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2003-3040
Record Dates: First submitted 2009-05-26; First posted 2009-05-27 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Stroke
Keywords: stroke cell therapy repair autologous
MeSH Terms: conditions — Stroke | interventions — SLC25A33 protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: placebo
- autologous mononuclear cells (Active Comparator): a single intravenous autologous bone marrow mononuclear cell transfusion
  Interventions: Biological: autologous bone marrow mononuclear cell transfusion
- autologous marrow stromal cells (Active Comparator): a single intravenous autologous marrow stromal cell transfusion
  Interventions: Biological: marrow stromal cells

INTERVENTIONS:
Biological: autologous bone marrow mononuclear cell transfusion — a single intravenous transfusion approximately 2 days after bone marrow aspiration, and 4 days after stroke onset; the full amount of autologous mononuclear cells derived from 30 cc of bone marrow
  Other Names: mononuclear cells
  Arms: autologous mononuclear cells
Biological: marrow stromal cells — a single intravenous transfusion approximately 21 days after bone marrow aspiration, and 23 days after stroke onset; the full amount of marrow stromal cells cultured over 21 days from 30 cc of bone marrow (expected to be approximately 1,000,000 cells/kg body weight)
  Other Names: mesenchymal stromal cells
  Arms: autologous marrow stromal cells
Drug: placebo — a single intravenous transfusion of saline, approximately 2-21 days after bone marrow aspiration, and 4-23 days after stroke onset; the full amount of mononuclear cells derived from 30 cc of bone marrow
  Arms: Placebo

SUMMARY:
This study will examine the safety of two different cellular therapies in the treatment of stroke.

DETAILED DESCRIPTION:
Stroke remains a leading cause of death and disability. A limited number of therapies, such as intravenous tissue plasminogen activator, have been approved to interrupt stroke in the early hours after symptom onset. Many patients are not able to benefit from these therapies, however, and so a need exists for development of new interventions to reduce disability after stroke. This study will be an early step towards this, and will examine the safety of two cell types, mononuclear cells and marrow stromal cells. In each case, the cells will be autologous, specifically being derived from the subject's own bone marrow.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke that is supratentorial in location and < 72 hours old between stroke onset and bone marrow aspiration
* No major pre-stroke disability
* NIH stroke scale score of 7-24
* Able to undergo bedside bone marrow aspiration
* Age 18-85 years, inclusive
* Reasonable likelihood of receiving standard physical, occupational and speech rehabilitation therapy

Exclusion Criteria:

* No major active hematological, immunological, or oncological diagnoses
* Pregnancy
* Lactating mothers
* At least 24 hours time of any thrombolytic therapy and time of bone marrow aspiration
* Allergy to penicillin or to fetal bovine serum
* Active, major co-existent neurological or psychiatric disease
* Infection with HIV, hepatitis B or C, or syphilis
* Any diagnosis that makes survival to 90 days post-stroke unlikely
* Participation in an experimental therapeutic clinical trial in the prior three months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
death | 90 days after stroke onset

SECONDARY OUTCOMES:
myocardial infarction | 90 days after stroke onset
pulmonary embolism | 90 days after stroke onset
ischemic stroke | 90 days after stroke onset
deep venous thrombosis | 90 days after stroke onset
other arterial or venous thrombosis | 90 days after stroke onset
Infection requiring IV antibiotics | 90 days after stroke onset

CONTACTS AND LOCATIONS:
Overall Officials: Steven C. Cramer, MD, MMSc, Principal Investigator — University of California, Irvine
Locations (1):
- UC Irvine Medical Center, Orange, California, United States

REFERENCES:
- [Background] Lane TA, Garls D, Mackintosh E, Kohli S, Cramer SC. Liquid storage of marrow stromal cells. Transfusion. 2009 Jul;49(7):1471-81. doi: 10.1111/j.1537-2995.2009.02138.x. Epub 2009 Mar 31. PMID 19389020